CLINICAL TRIAL: NCT05055895
Title: Association of Anticholinergic Burden With Onset of Delirium in Older Adults With Alzheimer Dementia: A Retrospective Cohort Study
Brief Title: Association of Anticholinergic Burden With Onset of Delirium in Older Adults With Alzheimer Dementia:
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bilal Katipoglu, Geriatric, Gulhane Training and Research Hospital
Other Study IDs: 2020-383
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Delirium; Anticholinergic Adverse Reaction; Alzheimer Disease
MeSH Terms: conditions — Delirium; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early onset deliryum on dementia: It was earlier than The median time of onset of delirium superimposed dementia
  Interventions: Drug: Anticholinergic burden
- Delirium on dementia (normal): It was equal or later than The median time of onset of delirium superimposed dementia
  Interventions: Drug: Anticholinergic burden

INTERVENTIONS:
Drug: Anticholinergic burden — The anticholinergic burden (ACB) was assessed using the Anticholinergic Burden Scale.
  Higher ACB was described as equal or higher than 1.

SUMMARY:
Drugs with anticholinergic properties are commonly prescribed to older persons despite growing evidence of their significant adverse effects. However, limited data are available concerning their contribution to time of onset of delirium. This study aimed to determine the potential association of higher anticholinergic burden to early-onset of delirium superimposed dementia in the older adult.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older and diagnosis or fellow-up of Alzhemier dementia in outpatient clinic.

Exclusion Criteria:

* The patients with a history of other than Alzhemier dementia or neurodegenerative disease (epilepsy, multiple sclerosis, Parkinson disease, etc.), terminal illness (malignancy, advanced organ failure) were excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All participiants enrolled from outpaitent clinic and underwent by comprehesive geriatric asssessment.
  Delirium and dementia status was assessed by the criteria of confusion assessment method (CAM) and DSM-4 or DSM-5 respectively.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Time onset of delirium superimposed dementia | 12 month
  First attack of delirium onset

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane training and research hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No